CLINICAL TRIAL: NCT03495167
Title: Multi-center, Open-label, Phase I Study of SyB C-1101 in Patients With Myelodysplastic Syndrome
Brief Title: Study of SyB C-1101 in Patients With Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SymBio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017001
Record Dates: First submitted 2017-11-17; First posted 2018-04-11 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SyB C-1101 (Experimental)
  Interventions: Drug: SyB C-1101

INTERVENTIONS:
Drug: SyB C-1101 — SyB C-1101 (rigosertib sodium) will be administered to two cohorts of patients; each receives either twice daily (560 mg before breakfast and 560 mg before dinner) or twice daily (840 mg before breakfast and 280 mg before dinner. SyB C-1101 will be administered orally twice daily for 21 consecutive days, followed by a 7-day observation period. The treatment period of 28 days (21 days of administration + 7 days of observation) constitutes 1 cycle.

SUMMARY:
To assess tolerability of SyB C-1101 when administered orally BID for 21 days followed by a 7-day observation period in patients with recurrent/relapsed or refractory myelodysplastic syndrome in order to determine a recommended dose (RD). To assess safety, efficacy and pharmacokinetics.

ELIGIBILITY:
Patients who meet all of the following criteria are eligible for enrollment in the study:

1. Histologically or cytologically diagnosed as myelodysplastic syndrome (MDS) according to WHO criteria or FAB classification. For patients with RAEB in transformation (RAEB-t), peripheral WBC is ≦25,000 /mm3 and the disease is stable for at least 4 weeks.
2. Classified as Intermediate-1, Intermediate-2 or High-risk, according to IPSS classification.
3. Patients with a history of previous treatment of the target disease (e.g., immunosuppressive therapy, protein anabolic steroids, and chemotherapy including azacitidine and lenalidomide) and meet one of the followings:

   * Patients who failed to achieve complete remission, partial remission, or hematologic improvement*
   * Patients experienced with recurrence/relapse after achieving complete remission, partial remission, or hematologic improvement*
   * Patients who were intolerable to the previous therapy *: The most recent assessment of the therapeutic effect based on "Clinical application and proposal for modification of the International Working Group (IWG) response criteria in myelodysplasia" (IWG2006 criteria)
4. Off all other treatment (including erythropoiesis stimulating agents) for MDS, for at least 4 weeks prior to enrollment and no carry-over (of antitumor effect) from previous treatment is expected as judged by Investigator. Transfusion is allowed, as clinically indicated.
5. Patients with expected survival of ≥3 months.
6. Patients aged 20 years or older (at the time of informed consent).
7. ECOG Performance Status (PS) of 0, 1 or 2
8. Patients with adequate major organ functions (including the heart, lungs, liver, and kidneys).

   * AST (GOT): ≤2.5 -fold the upper limit of normal range at each institution
   * ALT (GPT) : ≤2.5 -fold the upper limit of normal range at each institution
   * Total bilirubin: <2.0 mg/dL (except patients with Gilbert's disease or hemolysis)
   * Serum creatinine: <2.0 mg/dL
   * ECG: Absence of abnormal findings that require treatment
   * Echocardiography: Absence of abnormal findings that require treatment
9. The patient must sign an informed consent form indicating that s/he understands the purpose of and procedure required for the study and is willing to participate in the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-10-06 (Actual); Primary Completion 2019-05-28 (Actual); Study Completion 2019-05-28 (Actual)

PRIMARY OUTCOMES:
Identification of Dose-Limiting Toxicity (DLT) and Number of Patients with DLT in Each Cohort | Up to 2 years
  Based on the number of patients with DLT and administration dose in each cohort, recommended dosage will be defined for the following clinical phase.
  A DLT is defined as an adverse event that occurred during the Cycle 1, for which a causality with the investigational products (IP) cannot be ruled out and meets the following criteria.
  Criteria: ≥ Grade3 non-hematological toxicity (except pyrexia). However nausea, vomiting, diarrhea, stomatitis and esophagitis/dysphagia are excluded (≥ Grade 3 nausea, vomiting, and diarrhea persist for ≥ 48 hours and uncontrolled by antiemetic or antidiarrheal agents, and ≥ Grade 3 stomatitis and esophagitis/dysphagia lasting for ≥ 4 days are regarded as DLTs). ≥ Grade 2 pyrexia uncontrolled by antipyretic agents. However, in case pyrexia of ˃ 39°C occurred within 24 hours after administration of SyB C-1101 and its cause is unclear, it is deemed that the causality to the IP cannot be ruled out.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 2 years
  Calculate from the rate between number of patients occurred AE and number of patients received SyB C-1101.
Severity of adverse events | Up to 2 years
  Score as grade 1 to 5 according to criteria by CTCAE v4.0-JCOG.
Relationship of adverse events to SyB C-1101 | Up to 2 years
  Score as "related " or "not related".
Change of laboratory test values | Up to 2 years
  Number of patients with changes in laboratory values OR list each lab value separately (e.g.Hgb, Fe, Hct, etc.)
Overall hematologic response rate | Up to 2 years
  Calculate from the rate of patients scored as CR, PR or marrow CR according to IWG 2006 criteria.
Overall hematologic improvement rate | Up to 2 years
  Calculate from the rate of patients with hematologic improvement according to IWG 2006 criteria.
Overall cytogenetic response rate | Up to 2 years
  Calculate from the rate of patients scored as complete cytogeneic response or partial cytogenetic response according to IWG 2006 criteria.
Cmax | Up to 2 years
  Maximum plasma concentration
tmax | Up to 2 years
  Time to maximum plasma concentration
AUC | Up to 2 years
  Area under the plasma concentration curve
t 1/2 | Up to 2 years
  Half-life time

CONTACTS AND LOCATIONS:
Overall Officials: Katsuhisa Goto, Study Director — SymBio Pharmaceuticals
Locations (9):
- Japan (9):
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Maebashi, Gunma
  - Research Site, Sapporo, Hokkaido
  - Research Site, Kobe, Hyōgo
  - Research Site, Kurashiki, Okayama-ken
  - Research Site, Shinagawa, Tokyo
  - Research Site, Fukuoka
  - Research Site, Kumamoto
  - Research Site, Kyoto